CLINICAL TRIAL: NCT00086684
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Group Evaluation of the Efficacy and Tolerability of Two Different Doses of ELMIRON for the Treatment of Interstitial Cystitis
Brief Title: Effectiveness and Safety Study of Pentosan Polysulfate Sodium for the Treatment of Interstitial Cystitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim Analysis showed that study continuation was futile. No safety concerns were raised during the trial.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR004576; C-2002-036 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); NCT00399139 (obsolete NCT alias)
Record Dates: First submitted 2004-07-07; First posted 2004-07-09 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; Urinary Bladder Pain
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pentosan polysulfate sodium 100 mg once a day (Experimental): One 100 mg pentosan polysulfate sodium capsule in the morning and 1 matching placebo capsule in the afternoon and evening for 24 weeks
  Interventions: Drug: Pentosan polysulfate sodium 100 mg
- Pentosan polysulfate sodium 100 mg three times a day (Experimental): One 100 mg pentosan polysulfate sodium capsule 3 times a day (morning afternoon and evening) for 24 weeks
  Interventions: Drug: Pentosan polysulfate sodium 100 mg
- Placebo (Placebo Comparator): Placebo One placebo capsule 3 times a day (morning afternoon and evening) for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentosan polysulfate sodium 100 mg — One 100 mg pentosan polysulfate sodium capsule 3 times a day (morning, afternoon, and evening) for 24 weeks
  Arms: Pentosan polysulfate sodium 100 mg three times a day
Drug: Placebo — One placebo capsule 3 times a day (morning, afternoon and evening) for 24 weeks
  Arms: Placebo
Drug: Pentosan polysulfate sodium 100 mg — One 100 mg pentosan polysulfate sodium capsule in the morning, and 1 matching placebo capsule in the afternoon and evening for 24 weeks
  Arms: Pentosan polysulfate sodium 100 mg once a day

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of pentosan polysulfate sodium 100 mg once a day, pentosan polysulfate sodium 100 mg three times a day, and placebo for 24 weeks for the relief of bladder pain or discomfort associated with interstitial cystitis.

DETAILED DESCRIPTION:
The purpose of this multi-center, double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance), parallel group trial is to evaluate the effectiveness and safety of two doses of pentosan polysulfate sodium (100 mg once a day and 100 mg three times a day) versus placebo for 24 weeks for the relief of bladder pain or discomfort associated with interstitial cystitis. The hypothesis of the study is that there is no treatment difference in the proportion of responders at study endpoint (Week 24). Effectiveness will be assessed based on the reduction in the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) total score. Safety assessments include vital signs, laboratory tests, adverse events and physical exams. Patients will receive one of the following study treatments by mouth each day for 24 weeks: pentosan polysulfate sodium 100 mg once a day group - one pentosan polysulfate sodium 100 mg capsule in the morning, and one matching placebo capsule in the afternoon and evening; pentosan polysulfate sodium 100 mg capsule three times a day group - one pentosan polysulfate sodium 100 mg capsule in the morning, afternoon and evening; placebo group - one placebo capsule in the morning, afternoon and evening

ELIGIBILITY:
Inclusion Criteria:

* Must have a total score of 8 or greater on the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) and a score of > 0 on each of the 4 questions on the ICSI
* must have experienced bladder pain, urinary urgency and urinary frequency, each not related to a urinary tract infection, for at least 6 months prior to entry into the study
* must have averaged >= 10 voids per day (>=30 voids over 3 consecutive days) and averaged >= 1 void at night
* urine culture showing no evidence of urinary tract infection
* urine cytology showing no evidence of neoplastic cells

Exclusion Criteria:

* Scheduled for or use of intravesical therapy (eg, bladder distention, dimethyl sulfoxide) during or within 4 weeks prior to the study
* patients who have had cytoscopic evaluation within 4 weeks prior to the study
* patients who are currently (within last month) receiving other medications that may affect symptoms of interstitial cystitis (ie, antidepressants, antihistamines, antispasmodics, anticholinergics)
* patients who are chronic users of Schedule II narcotics or who are using any scheduled narcotics at the time of study entry
* patients taking coumadin, anticoagulants, heparin, or thrombolytic agents such as tissue plasminogen activator and streptokinase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2003-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (65):
- United States (52):
  - Birmingham, Alabama
  - Homewood, Alabama
  - Anchorage, Alaska
  - San Bernardino, California
  - San Carlos, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Longmont, Colorado
  - Wheat Ridge, Colorado
  - Newington, Connecticut
  - Norwalk, Connecticut
  - Celebration, Florida
  - Longwood, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Trinity, Florida
  - Venice, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Centralia, Illinois
  - Evanston, Illinois
  - Peoria, Illinois
  - Jeffersonville, Indiana
  - Dearborn, Michigan
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - St Louis, Missouri
  - Henderson, Nevada
  - West Orange, New Jersey
  - Albany, New York
  - Charlotte, North Carolina
  - Concord, North Carolina
  - Winston-Salem, North Carolina
  - Lima, Ohio
  - Ponca City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Mountlake Terrace, Washington
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (13):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Surrey, British Columbia
  - Victoria, British Columbia
  - Fredericton, New Brunswick
  - Halifax, Nova Scotia
  - Kentville, Nova Scotia
  - Barrie, Ontario
  - Burlington, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred and sixty-nine patients enrolled in this study. One patient did not take any study drug. Therefore, only 368 patients were included in the primary analysis dataset.
Groups:
- Pentosan Polysulfate Sodium (ELMIRON) 100MG QD: One 100 mg pentosan polysulfate sodium capsule QD (once daily)
- Pentosan Polysulfate Sodium (ELMIRON) 100MG TID: One 100 mg pentosan polysulfate sodium capsule TID (three times a day)
Period: Overall Study
Arm/Group | PLACEBO | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID
Started | 118 | 129 | 122
Completed | 63 | 74 | 69
Not Completed | 55 | 55 | 53
Not completed — Adverse Event | 12 | 17 | 14
Not completed — Lack of Efficacy | 6 | 6 | 5
Not completed — Lost to Follow-up | 15 | 8 | 10
Not completed — Protocol Violation | 8 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 10
Not completed — NONCOMPLIANCE | 5 | 7 | 6
Not completed — STUDY TERMINATED BY SPONSOR | 0 | 1 | 0
Not completed — WITHDRAWAL OF CONSENT | 5 | 7 | 5
Not completed — Other | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID | Total
Number analyzed (Participants) | 118 | 129 | 122 | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 2
  Between 18 and 65 years | 103 | 108 | 109 | 320
  >=65 years | 14 | 20 | 13 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (14.58) | 45.6 (15.68) | 42.7 (15.71) | 44.3 (15.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 119 | 113 | 333
  Male | 17 | 10 | 9 | 36
AgeCategorical [Number; unit: participants]
  <18 YEARS | 0 | 0 | 0 | 0
  18-<64 YEARS | 104 | 109 | 109 | 322
  65-<74 YEARS | 10 | 17 | 11 | 38
  >=75 YEARS | 4 | 3 | 2 | 9
Baseline BMI [Mean (Standard Deviation); unit: kg/cm2] | 27 (6.50) | 26.8 (9.42) | 27.1 (11.02) | 26.9 (9.18)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders Defined as Having at Least a 30% Reduction in the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) From Baseline to Study Endpoint
Description: The ICSI is a four-item self-administered instrument developed for the evaluation and management of patients with interstitial cystitis. The index measures the presence and extent of symptoms including urinary urgency, urinary frequency, nocturia and pain/burning in the bladder. Each question in the ICSI is on a 0-5 scale, where each answer is given a specific rating. The sum of the individual question ratings is the score for the ICSI. The range of the test is a score of 0 to 20. A lower score indicates a better condition.
Time Frame: Baseline to Week 24
Population: Intent-to-Treat (ITT) Analysis set
Measure: Number; unit: participants
Arm/Group | PLACEBO | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID
Number analyzed (Participants) | 118 | 128 | 122
participants | 48 | 51 | 52

2. Secondary Outcome: Number of Responders Defined as Having at Least a Four Point Reduction in the O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) From Baseline to Study Endpoint
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: Intent-to-Treat (ITT) Analysis set
Measure: Number; unit: participants
Arm/Group | PLACEBO | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID
Number analyzed (Participants) | 118 | 128 | 122
participants | 55 | 55 | 60

ADVERSE EVENTS:
Arm/Group | PLACEBO | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID
Serious Adverse Events (participants affected / at risk) | 4/118 | 4/128 | 0/122
Other Adverse Events (participants affected / at risk) | 95/118 | 107/128 | 97/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=118) | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD (N=128) | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID (N=122)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder Cholesterolosis (Hepatobiliary disorders) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Homicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Renal Mass (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=118) | Pentosan Polysulfate Sodium (ELMIRON) 100MG QD (N=128) | Pentosan Polysulfate Sodium (ELMIRON) 100MG TID (N=122)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 1
Stargardt's Disease (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0
Motion Sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Conjunctival Hyperaemia (Eye disorders) | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1
Macular Degeneration (Eye disorders) | 0 | 1 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 2
Visual Acuity Reduced (Eye disorders) | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 3 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 3
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 13 | 6
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 2 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 19 | 12
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1
Tooth Impacted (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 10 | 4
Asthenia (General disorders) | 0 | 2 | 0
Chest Discomfort (General disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 2
Malaise (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 1 | 2
Pain (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Suprapubic Pain (General disorders) | 0 | 1 | 0
Tenderness (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Seasonal Allergy (Immune system disorders) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Ear Infection (Infections and infestations) | 2 | 2 | 1
Eye Infection (Infections and infestations) | 0 | 2 | 0
Fungal Infection (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Gastroenteritis Viral (Infections and infestations) | 2 | 1 | 0
Gingival Infection (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 3
Localised Infection (Infections and infestations) | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1
Otitis Externa (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pharyngitis Streptococcal (Infections and infestations) | 2 | 4 | 1
Purulent Discharge (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 2
Tooth Abscess (Infections and infestations) | 0 | 0 | 3
Tooth Infection (Infections and infestations) | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 9 | 8
Vaginitis Bacterial (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1 | 3
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Cholesterol Increased (Investigations) | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 2 | 2 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 1
Blood Urine Present (Investigations) | 0 | 1 | 0
Cardiac Murmur (Investigations) | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Monocyte Count Increased (Investigations) | 0 | 0 | 1
Prothrombin Time Prolonged (Investigations) | 0 | 0 | 1
Smear Cervix Abnormal (Investigations) | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 5
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mycosis Fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 8
Headache (Nervous system disorders) | 16 | 16 | 14
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 2 | 5
Lethargy (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 2 | 2 | 1
Migraine with Aura (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0 | 0
Sinus Headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Libido Decreased (Psychiatric disorders) | 1 | 1 | 0
Mood Swings (Psychiatric disorders) | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 1
Bladder Discomfort (Renal and urinary disorders) | 0 | 1 | 0
Bladder Pain (Renal and urinary disorders) | 38 | 35 | 47
Bladder Prolapse (Renal and urinary disorders) | 0 | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 1 | 1
Cystitis Interstitial (Renal and urinary disorders) | 11 | 19 | 9
Dysuria (Renal and urinary disorders) | 2 | 2 | 3
Haematuria (Renal and urinary disorders) | 1 | 2 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Urethral Pain (Renal and urinary disorders) | 1 | 0 | 0
Urethral Ulcer (Renal and urinary disorders) | 0 | 1 | 0
Atrophic Vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 3 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Vaginal Odour (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Influenza (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 14 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 5
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Heat Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Idiopathic Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No